CLINICAL TRIAL: NCT05082597
Title: Clinical Outcome of Extracorporeal Shock Wave Therapy in Patient With Axillary Web Syndrome-A Pilot Study
Brief Title: Clinical Outcome of Extracorporeal Shock Wave Therapy in Patient With Axillary Web Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF21163B
Record Dates: First submitted 2021-09-24; First posted 2021-10-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Axillary Web Syndrome; Breast Cancer; Lymphedema; Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ESWT (Experimental): Receive low energy extracorporeal shock wave therapy
  Interventions: Device: Low energy ESWT

INTERVENTIONS:
Device: Low energy ESWT — Therapeutic sessions: 4(once a week, for 4 weeks) Total dosage: 2500 shoots over axillary cord lesion (1000 over most fibrotic area, 500 over upper arm, 500 over forearm, 500 over other area) Energy: 0.056-0.065mJ/mm2

SUMMARY:
Axillary web syndrome(AWS) is common complication of breast cancer surgery. Overall, AWS affects more than a half of the patient receiving axillary lymph node dissection. The symptoms of AWS include pain, limited function and range of motion. Geater risk of secondary lymphedema was found if the patient developed AWS during the first postoperative year.

ESWT was used for treating myofascial pain for decades. Low energy ESWT combined with complex decongestive therapy had a benefit on shoulder joint ROM and skin thickness improvement in patients with BCRL in recently studies. Investigators wonder if ESWT can also be applied to patients with axillary web syndrome for increasing ROM and relieving pain.

The aim of this study was to evaluate the therapeutic effects of low energy ESWT in patients with axillary web syndrome.

DETAILED DESCRIPTION:
Although the anticipated enrollment was 30 participants, the study was completed with 20 participants due to early attainment of statistical significance and recruitment feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Axillary web syndrome patient
2. Unilateral breast cancer and received related operation(mastectomy/ALND/SLND)
3. Completion of beast related chemotherapy or radiotherapy
4. Age with 20-65 years old

Exclusion Criteria:

1. Ongoing metastasis or recurrence of the breast cancer
2. Other cancer history
3. Lymphatic transplantation or reconstruction
4. Wound, infection or trauma over affected arm
5. Coagulopathy or poor circulation
6. Pregnancy
7. Oral anticoagulant using

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Shoulder range of motion | 2 months
  Flexion, extension, external rotation, internal rotation, abduction over upper limbs
Pain score | 2 months
  Visual Analogue Scale (0-10 points, higher score represented higher degree of pain)

SECONDARY OUTCOMES:
Muscle strength | 2 months
  Muscle strength of upper limb measured by ergometer
Upper limb functional score | 2 months
  quick Disabilities of the Arm, Shoulder and Hand Score(qDASH) (0-100 points, higher score indicated higher level of upper limb impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Lin Tsai, MD, Study Chair — Department of Physical Medicine and Rehabilitation
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No